CLINICAL TRIAL: NCT02722629
Title: Prevalence of Respiratory Aspiration in Patients With COPD: Cross-sectional Study
Brief Title: Prevalence of Respiratory Aspiration in Patients With COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Collaborators: ATS MECOR (Methods in Epidemiologic, Clinical and Operations Research) Latin America program - Faculty Team (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2671
Record Dates: First submitted 2016-03-09; First posted 2016-03-30 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-03

CONDITIONS: COPD
Keywords: COPD; Respiratory Aspiration; COPD acute exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aspiration in COPD patients (Experimental): All COPD patient will be evaluated systematically by FEESST (Flexible Endoscopic Evaluation of Swallowing with Sensory Testing) with direct evaluation of aspiration by direct observation.
  Interventions: Procedure: FEESST

INTERVENTIONS:
Procedure: FEESST — Flexible Endoscopic Evaluation of Swallowing with Sensory Testing

SUMMARY:
The aim of the study is to estimate the prevalence of respiratory aspiration in patients with COPD, in a tertiary hospital of Buenos Aires.

DETAILED DESCRIPTION:
Primary objective To estimate the prevalence of respiratory aspiration in patients with COPD, in a tertiary hospital of Buenos Aires.

Secondary objective

1. To assess the association between the presence of aspiration and the usual degree of dyspnea in patients with COPD.
2. To assess the association between the presence of aspiration and the amount of regular annual exacerbations in patients with COPD.
3. To evaluate the association between the presence of aspiration and degree of severity according to GOLD criteria in patients with COPD.
4. Compare the estimated aspiration in COPD patients with known prevalence of pulmonary aspiration in the general population in the same age patient prevalence

Patients will be recruited consecutively in the outpatient clinic of Pulmonology and Medical Clinic, where a first encounter with the patient will be agreed. Additionally, the investigators will cite patients identified as COPD in the Electronic Medical Records.

During the first meeting the informed consent process to enter the protocol will take place, then the same baseline characteristics of the patient is taken into an online form. Finally given a shift within 15 days after the first meeting for the FEEST, and if the patient did not have a spirometry over the past year to update a new turn. Both studies will be conducted without any cost.

In patients with impaired swallowing or aspiration presence is detected, we will inform the doctor to assess the need for additional studies. In turn, the patients will be referred to speech therapy services for rehabilitation of swallowing.

ELIGIBILITY:
Inclusion Criteria

- Patients over 64 years diagnosed with chronic obstructive pulmonary disease guide GOLD criteria (FEV1 / FVC ratio post bronchodilator <0.70)

Exclusion Criteria

* Refusal to participate or to process oral informed consent
* Contraindication for the FEESST (history of vasovagal episodes, bilateral nasal obstruction, impaired homeostasis or frequent bleeding, dyskinesia, maxillofacial trauma or recent neck).
* Impaired understanding or cognition that hinder the consent or performing diagnostic tests required.
* Diagnosis of neurodegenerative disease associated with swallowing disorders known: Parkinson, stroke with neurologic sequelae.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Presence of any consistence Airway Aspiration | Baseline (Time 0)
  Direct observation of any consistence food (liquid/semisolid/solid) penetration or aspiration by direct inspection with Flexible Endoscopic Evaluation of Swallowing with Sensory Testing.
  There is no follow-up period as this is a prevalence study. All measurements will be done at time 0. The only experimental feature (according to ClinicalTrials.gov definitions) is that we use FEEST to detect evidence of airway aspiration and this is not a routine examination in COPD patients.

SECONDARY OUTCOMES:
Aspiration Risk | Baseline (Time 0)
  Direct observation of indirect signs of high risk for aspiration with Flexible Endoscopic Evaluation of Swallowing with Sensory Testing.
  There is no follow-up period as this is a prevalence study. All measurements will be done at time 0. The only experimental feature (according to ClinicalTrials.gov definitions) is that we use FEEST to detect evidence of airway aspiration and this is not a routine examination in COPD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Hernan Benito, MD, Principal Investigator — Hospital Italiano de Buenos Aires; Diego h Giunta, MD, Principal Investigator — Hospital Italiano de Buenos Aires; Fernando Warley, MD, Principal Investigator — Hospital Italiano de Buenos Aires; Bruno Ferreyro, MD, Principal Investigator — Hospital Italiano de Buenos Aires; Federico Sala, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Peron 4190, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Lopez AD, Shibuya K, Rao C, Mathers CD, Hansell AL, Held LS, Schmid V, Buist S. Chronic obstructive pulmonary disease: current burden and future projections. Eur Respir J. 2006 Feb;27(2):397-412. doi: 10.1183/09031936.06.00025805. No abstract available. PMID 16452599
- [Result] Ciapponi A, Alison L, Agustina M, Demian G, Silvana C, Edgardo S. The epidemiology and burden of COPD in Latin America and the Caribbean: systematic review and meta-analysis. COPD. 2014 Jun;11(3):339-50. doi: 10.3109/15412555.2013.836479. Epub 2013 Oct 10. PMID 24111903
- [Result] Steidl E, Ribeiro CS, Goncalves BF, Fernandes N, Antunes V, Mancopes R. Relationship between Dysphagia and Exacerbations in Chronic Obstructive Pulmonary Disease: A Literature Review. Int Arch Otorhinolaryngol. 2015 Jan;19(1):74-9. doi: 10.1055/s-0034-1376430. Epub 2014 Nov 6. PMID 25992155
- [Result] Macri MR, Marques JM, Santos RS, Furkim AM, Melek I, Rispoli D, de Alencar Nunes MC. Clinical and fiberoptic endoscopic assessment of swallowing in patients with chronic obstructive pulmonary disease. Int Arch Otorhinolaryngol. 2013 Jul;17(3):274-8. doi: 10.7162/S1809-97772013000300007. PMID 26106452
- [Result] Yamauchi Y, Yasunaga H, Matsui H, Hasegawa W, Jo T, Takami K, Fushimi K, Nagase T. Comparison of clinical characteristics and outcomes between aspiration pneumonia and community-acquired pneumonia in patients with chronic obstructive pulmonary disease. BMC Pulm Med. 2015 Jul 8;15:69. doi: 10.1186/s12890-015-0064-5. PMID 26152178